CLINICAL TRIAL: NCT07207174
Title: Dual-Language Brief Mindfulness-Oriented Recovery Enhancement (B-MORE) vs Brief Cognitive-Behavioral Therapy (B-CBT) for Chronic Pain
Brief Title: Brief Mindfulness-Oriented Recovery Enhancement vs Brief Cognitive-Behavioral Therapy for Chronic Pain
Acronym: B-MORE v B-CBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Assistant Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00006512
Record Dates: First submitted 2025-09-17; First posted 2025-10-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain
Keywords: Chronic pain; Spanish-language intervention; Mindfulness; Cognitive-behavioral Therapy; Brief intervention
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Behavioral Intervention #1 (Experimental): Brief Mindfulness Oriented Recovery Enhancement (B-MORE)
  Interventions: Behavioral: Brief Mindfulness Oriented Recovery Enhancement
- Brief Behavioral Intervention #2 (Experimental): Brief Cognitive-Behavioral Therapy (B-CBT)
  Interventions: Behavioral: Brief Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Brief Mindfulness Oriented Recovery Enhancement — B-MORE is a 2-hour adaptation of the traditional MORE program.
  Arms: Brief Behavioral Intervention #1
Behavioral: Brief Cognitive-Behavioral Therapy — B-CBT is a 2-hour adaptation of a traditional 8-week CBT for Chronic Pain manual.
  Arms: Brief Behavioral Intervention #2

SUMMARY:
This randomized controlled trial aims to test both English and Spanish versions of two, benign behavioral interventions for adults with chronic pain -- 1) Brief Mindfulness-Oriented Recovery Enhancement (B-MORE), and 2) Brief Cognitive- Behavioral Therapy (B-CBT).

ELIGIBILITY:
Inclusion Criteria:

* Having a chronic pain condition
* Average pain of > 3 in the last week
* Willingness to engage with study assessments and interventions
* Understanding English or Spanish instructions fluently
* Age 18 and above.

Exclusion Criteria:

* Unable to consent because of physical or mental incapacity
* Have previous, formal mindfulness or CBT training (e.g., MBSR)
* Have pain from a current cancer diagnosis
* Unstable illness that may interfere with treatment
* Had surgery within the previous three months
* Had pain relieving injections, such as cortisone or hyaluronate, within the previous three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2027-09-22 (Estimated); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
Program Feasibility | At the first treatment session [1 hour] and the final treatment session [1 hour]
  Feasibility will be assessed by intervention adherence rates (percentage of treatment sessions completed).
Treatment Acceptability | Upon completion of the final treatment session [1 hour]
  Treatment acceptability will be assessed by an adaptation of the Theoretical Framework of Acceptability scale (TFA).

SECONDARY OUTCOMES:
Chronic Pain Symptoms | Baseline and 2, 6, and 12-week post-treatment follow-ups
  Chronic Pain Symptoms will be measured via the Pain, Enjoyment, and General Activity scale (PEG-3).
Depressive Symptoms | Baseline and 2, 6, and 12-week post-treatment follow-ups
  Depressive Symptoms will be measured with the Patient Health Questionnaire (PHQ-2).
Anxiety Symptoms | Baseline and 2, 6, and 12-week post-treatment follow-ups
  Anxiety Symptoms will be measured with the Generalized Anxiety Disorder questionnaire (GAD-2).
Wellbeing | Baseline and 2, 6, and 12-week post-treatment follow-ups
  Wellbeing will be measured with the World Health Organization Wellbeing Index (WHO-5).
Pain Catastrophizing | Baseline and 2, 6, and 12-week post-treatment follow-ups
  Pain Catastrophizing will be measured with a validated 4-item adaptation of the Pain Catastrophizing scale (PCS-4).

OTHER OUTCOMES:
Credibility/Expectancy | Immediately upon completion of the first treatment session
  Treatment Credibility/Expectancy will be measured with an adaptation of the Credibility and Expectancy Questionnaire (CEQ).
Mindful Reappraisal of Pain Sensations | Baseline and 2, 6, and 12-week post-treatment follow-ups
  Mindful Reappraisal of Pain Sensations will be measured with the Mindful Reappraisal of Pain Sensations scale (MRPS-9).
Trait Decentering | Baseline and 2, 6, and 12-week post-treatment follow-ups
  Trait Decentering will be measured with the 3-item Metacognitive Processes of Decentering Scale
Trait Self-Transcendence | Baseline, and at 2, 6, and 12-week post-treatment follow-ups
  Trait Self-Transcendence will be measured with the 3-item Nondual Awareness Dimensional Scale
Acute Pain Intensity/Unpleasantness | Immediately before and after treatment sessions #1 (first) and #2 (last)
  Acute Pain Intensity/Unpleasantness will be assessed with a 0-10 Numeric Rating Scale before and after each treatment session.
Acute Anxiety | Immediately before and after treatment sessions #1 (first) and #2 (last)
  Acute Anxiety will be assessed with a 0-10 numeric rating scale before and after each treatment session.
State Decentering | Immediately before and after treatment sessions #1 (first) and #2 (last)
  State Decentering will be measured with the 3-item questionnaire - Metacognitive Processes of Decentering Scale (MPoDS)
State Self-Transcendence | Immediately before and after treatment sessions #1 (first) and #2 (last)
  State Self-Transcendence will be measured with the 3-item Nondual Awareness Dimensional Assessment (NADA).
Optional Neuroimaging Session: EEG | After study completion at the 12-week post-treatment follow-up.
  Spanish-speaking participants will be invited to participate in an optional neuroimaging session. EEG will be collected and analyzed during a baseline period and a mindfulness meditation task.
Optional Neuroimaging Session: fNIRS | After study completion at the 12-week post-treatment follow-up.
  Spanish-speaking participants will be invited to participate in an optional neuroimaging session. Functional Near-Infrared Spectroscopy (fNIRS) will be collected and analyzed during a baseline period and a mindfulness meditation task.
Acute Pain Medication Desire | Treatment session #1 [1 hour] and treatment session #2 [1 hour]
  Acute Pain Medication Desire will be assessed via a 0-10 numeric rating scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Building B, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, SAP, ICF, and de-identified IPD will be shared with qualified individuals upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: It will be available from study end up to 5 years afterwards.
Access Criteria: Any qualified individual may request the above-mentioned IPD and supporting information from the research team. Research team will provide the above via secure individual correspondence.